CLINICAL TRIAL: NCT03638115
Title: Clinical Investigation of the Safety & Effectiveness of the VaSecure 018 Drug Coated PTA Balloon Catheter in the Treatment of Patients With Chronic Limb Threatening Ischemia (CLTI) Involving Below-the-Knee (BTK) Arteries
Brief Title: The VaSecure BTK Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vascuros Medical Pte Ltd (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEC-BTK-001
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VaSecure™ Drug Coated PTA Balloon Catheter (Experimental)
  Interventions: Device: VaSecure™

INTERVENTIONS:
Device: VaSecure™ — Drug Coated PTA Balloon Catheter

SUMMARY:
To assess the safety and performance of the VaSecure drug-coated PTA balloon catheter in the treatment of patients with Chronic Limb Threatening Ischemia (CLTI) of the lower limb below the knee (BTK)

DETAILED DESCRIPTION:
The VaSecure Drug Coated PTA Balloon Catheter is indicated for percutaneous transluminal angioplasty (PTA), after predilatation, of de novo lesions in the peripheral vasculature of the lower limb with reference vessel diameters of 2-4 mm.

The study will include patients with lesions located in the infrapopliteal arteries diagnosed with CLTI of Rutherford categories 3-5. A maximum number of 46 patients will be enrolled in this clinical investigation in 7 sites in Europe and 2 in Singapore.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to participating in the clinical investigation, e.g. patients are mentally able to understand the aim of the clinical investigation.
2. Has a documented diagnosis of CLTI of Rutherford category 3-5.
3. The target lesion must be de novo.
4. Life expectancy is >1 year, in the investigator's opinion.
5. For women: menopausal or under active birth control.
6. Patient must agree not to participate in any other clinical trial during 12 month follow-up period.

   Visual angiographic inclusion criteria
7. Reference vessel(s) diameter is between 2mm-4mm. Each lesion in one or maximum two of the infrapopliteal arteries NOT extending beyond the ankle joint. Target lesion(s) consisting of a single solitary or series of multiple adjacent lesions (all less than 30 mm apart) in a single tibial vessel with a diameter stenosis ≥70% and a cumulative length of ≥50 mm to ≤250 mm. If there are two target lesions they will be separated for ≥3 cm and will be named from proximal to distal. Target lesion must be a tibial vessel (excluding popliteal artery) branching from popliteal artery.

Exclusion Criteria:

1. Breastfeeding or pregnant woman.
2. Severe concentric calcification, documented by angiography using the COMPLIANCE360-Score (This scoring system takes into account both the arc of calcium (< or > 180º) and percent of lesion length (< or > 50%) as judged by fluoroscopy.) that could not be fully expanded by predilatation balloon and documented by angiography. Valid record up to 30 days before screening.
3. Patients with major amputations that have already been performed or are planned, either on the target leg or on the contralateral side. .
4. History of stroke within 3 months.
5. History of myocardial infarction, thrombolysis or angina within 30 days prior to index procedure.
6. Renal failure or chronic kidney disease with estimated Glomerular Filtration Rate (eGFR) ≤30 mL/min per 1.73 m2 (or serum creatinine ≥2.5 mg/dL within 30 days of index procedure or treated with dialysis).
7. Diagnosed active untreated systemic infection or uncontrolled coagulopathy within 14 days prior to index procedure.
8. Co-morbid conditions limiting life expectancy to <12 months.
9. Hemorrhagic diathesis or another disorder such as gastrointestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anticoagulation therapy.
10. Known allergy to paclitaxel or paclitaxel-related compounds or contrast media that cannot be adequately managed with pre- and post-procedure medication.
11. Is currently participating in an investigational drug or other investigational device study or previously enrolled in this study.
12. Is unlikely to comply with the follow up schedule.
13. Has uncontrolled ulcer wound infection.
14. Is unwilling to comply with a concurrent ulcer wound therapy.
15. Has an allergy to acetylsalicylic acid, prasugrel, ticagrelol, and clopidogrel (Plavix®).
16. Use of atherectomy in proximal vessels or TL. However, the use of scoring/cutting balloons in the TL is allowed.

    Angiographic exclusion criteria
17. Lesions that cannot be successfully predilated to achieve a residual stenosis of <50% by visual estimate.
18. Severe dissection post dilatation resulting in a flow limiting lesion.
19. Thrombus in the target vessel documented by angiography.
20. Aneurysm in the target vessel(s).
21. Treatment of the contralateral limb during the same index procedure or within 30 days post-index procedure in order to avoid confounding complications.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from a composite endpoint of Major adverse limb event (MALE) and procedure-related mortality. | 30 days
  Major adverse limb event is defined as the composite of either major amputation or major re-intervention through 30 days of the index procedure.

SECONDARY OUTCOMES:
Procedure success rate | Index procedure or 1 day post index procedure
  Composite of technical success defined as successful vascular access and completion of the endovascular procedure as well as immediate morphological success with <30% residual reduction in diameter as assessed by QVA and Device success defined as exact deployment of the device according to the Instructions For Use (IFU) as documented by suitable imaging means
Incidence of all Adverse Events (AEs) | 30 days, and 3, 6, 9 and 12 months
  All AEs will be characterized by severity, relatedness, outcome and treatment
Freedom from major target limb amputation | 3, 6, 9 and 12 months
  Rates of amputation of the lower limb above 1 cm from the ankle mortice/joint upwards
Freedom from clinically-driven target lesion revascularization (cd-TLR) and target vessel revascularization (TVR) | 3, 6, 9 and 12 months
  Clinically-driven TLR is defined by core lab confirmation of restenosis ≥70% in the target lesion with wound persistence, new wounds or re-occurence of ischemic rest pain
Late Lumen Loss (LLL) of the target lesion | 6 months
  As measured by QVA
Angiographic Restenosis | 6 months
  Defined as ≥70% diameter stenosis on 2-view angiography by visual estimate
Angiographic Restenotic Burden | 6 months
  Defined as the percentage of length of stenosis/occlusion ≥70% on 2-view angiography by visual estimate in mm, divided by the total length of the lesion in mm
Freedom from occlusion (FFO) without cd-TLR on Duplex ultrasound | 3, 6 and 9 months
  Defined as presence of flow on colour doppler of the target lesion
Haemodynamic microvascular performance | Baseline, 3, 6 and 12 months
  As measured by transcutaneous oxygen (TcpO2)
Haemodynamic microvascular performance | Baseline, 6 and 12 months
  As measured by Ankle-Brachial-Index (ABI).
Wound healing rate | 30 days, 3, 6, 9 and 12 months.
  Defined as healed or not, if not, improving, stagnant or worsening
Rutherford status | 3, 6, 9 and 12 months
  Change in Rutherford classification as assessed by the investigator
Clinical Improvement (combined endpoint) in amputation free, cd-TLR free, surviving patients | 3, 6, 9 and 12 months
  Specified as an improvement shift in the Rutherford classification of one class.
Limb salvage | 6 and 12 months
  Defined as preservation of a functional foot without the need for a leg prosthesis
Amputation-free survival | 6 and 12 months
  Defined as composite endpoint of mortality and amputation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Universitaets-Herzzentrum Freiburg - Bad Krozingen GmbH
Locations (7):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Regionaal Ziekenhuis Heilig Hart, Tienen
- Germany (3):
  - Klinikum Hoschsauerland, Arnsberg
  - Universitaetsklinikum Muenster, Münster
  - Regiomed Kliniken Sonneberg, Sonneberg
- Singapore (2):
  - Changi General Hospital, Singapore
  - National University Hospital, Singapore